CLINICAL TRIAL: NCT00653081
Title: Supervised Exercises Compared With Radial Extracorporal Shock Wave Therapy (rESWT) in Patients With Subacromial Impingement Syndrome: A Single Blind Clinical Randomized Study
Brief Title: Supervised Exercises Compared With Radial Extracorporal Shock Wave Therapy (rESWT) in Patients With SIS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: South Eastern Area Health Service (Other); University of Oslo (Other)
Responsible Party: University of Oslo, South Eastern Area Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VT; rESWT
Record Dates: First submitted 2008-01-07; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2007-01

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Supervised Exercises; Radial Shock Wave Therapy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Supervised Exercises performed at ulleval Hospital for patients with shoulder pain. Dosage: 45 minutes each time, max 2-3 times a week in max 12 weeks
  Interventions: Procedure: Physical therapy method called Supervised Exercises
- B (Active Comparator): Radial Shock Wave therapy performed at ulleval Hospital, once a week, 4-6 times, 3-5 points each time.
  Interventions: Procedure: Radial Extracorporeal Shockwave Therapy

INTERVENTIONS:
Procedure: Physical therapy method called Supervised Exercises — Performed at ullevaal Hospital, 45 min each time, 2-3 times pr week in max 12 weeks
  Arms: A
Procedure: Radial Extracorporeal Shockwave Therapy — Radial Shock Wave therapy performed at ulleval Hospital, once a week, 4-6 times, 3-5 points each time.
  Arms: B

SUMMARY:
The purpose of this study is to compare Supervised Exercises with another non-operative frequently used treatment, Radial Extracorporeal Shockwave Therapy (rESWT), for patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain is, in succession to back, neck, and knee, the fourth most frequently localized musculoskeletal pain reported by patients to general practitioners and physical therapists. A majority of shoulder complaints lasts for more than three months and become chronic. Few of the different interventions for rehabilitation of chronic shoulder pain, have documented effect. Patients with shoulder pain are associated with significant disability and loss of quality of life which interfere with activities related to daily living.

Supervised exercises, a treatment method which has been compared to surgery and placebo laser, is one that has documented effect for both short (6 months) and long time (2½ years). The purpose of this study was to compare Supervised Exercises with another non-operative common used treatment method for these patients, radial Extracorporeal Shockwave Therapy (rESWT).

The study is designed as a randomised, single blind clinical controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial shoulder pain lasting for at least three months and age between 18 and 70 years.
* Dysfunction or pain on abduction
* Had a normal passive glenohumeral range of movement
* Pain during two of three isometric tests (abduction, external- or internal rotation at 0º or 30º)
* Positive Hawkins-Kennedys test.

Exclusion Criteria:

* Shoulder pain bilateral (both shoulders required treatment)
* Earlier operated in affected shoulder
* Had multidirectional instability
* Had the cervical syndrome
* Rheumatoid arthritis
* Clinical and radiological findings indicating glenohumeral - or acromioclavicular joint pathology
* Not able to understand spoken or written Norwegian
* Considerable emotional distress
* Needed anticoagulant medicine
* Being pregnant
* Had had Shock Wave Therapy or Supervised Exercises before.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline, 6 weeks, 12 weeks, 18 weeks and 12 months

SECONDARY OUTCOMES:
Pain intensity labelled "no pain" and "severe pain" at its extremes, are measured on nine point scales for activity and rest during last week. | Baseline, 6 weeks, 12 weeks, 18 weeks and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kaia Engebretsen, PhD, Principal Investigator — Dep of Physical Medicine and rehabilitation, Ullevaal University Hospital, Oslo, Norway
Locations (1):
- Department for physical medicine and rehabilitation, Ullevaal University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Engebretsen K, Grotle M, Bautz-Holter E, Ekeberg OM, Juel NG, Brox JI. Supervised exercises compared with radial extracorporeal shock-wave therapy for subacromial shoulder pain: 1-year results of a single-blind randomized controlled trial. Phys Ther. 2011 Jan;91(1):37-47. doi: 10.2522/ptj.20090338. Epub 2010 Nov 18. PMID 21088117
- [Derived] Engebretsen K, Grotle M, Bautz-Holter E, Ekeberg OM, Brox JI. Predictors of shoulder pain and disability index (SPADI) and work status after 1 year in patients with subacromial shoulder pain. BMC Musculoskelet Disord. 2010 Sep 23;11:218. doi: 10.1186/1471-2474-11-218. PMID 20863369
- [Derived] Engebretsen K, Grotle M, Bautz-Holter E, Sandvik L, Juel NG, Ekeberg OM, Brox JI. Radial extracorporeal shockwave treatment compared with supervised exercises in patients with subacromial pain syndrome: single blind randomised study. BMJ. 2009 Sep 15;339:b3360. doi: 10.1136/bmj.b3360. PMID 19755551